CLINICAL TRIAL: NCT02607150
Title: Changes in Cerebral Oxygenation During the Administration of Cell Saver Blood and Allogeneic Blood
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chairman, Department of Anesthesiology and Pain Medicine, Nationwide Children's Hospital
Other Study IDs: IRB14-00889
Record Dates: First submitted 2015-11-16; First posted 2015-11-17 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Idiopathic Scoliosis; Transfusion Reaction
Keywords: Spinal Fusion; Cerebral Oxygenation; Blood Transfusion
MeSH Terms: conditions — Transfusion Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Cerebral Oxygenation Changes — Monitor cerebral oxygenation changes in patients receiving blood transfusions who are undergoing spinal fusion surgery.

SUMMARY:
A prospective study designed to evaluate changes in tissue and cerebral oxygenation before and following administration of blood for patients undergoing spinal surgery.

Red blood transfusions (autologous and allogeneic) are indicated to improve oxygen delivery to the tissues and hence tissue oxygenation. Despite the presumed efficacy, there are limited data to demonstrate changes in tissue oxygenation with the administration of blood. Furthermore, the administration of both autologous blood from cell saver and allogeneic blood can be associated with both acute and long-term deleterious physiologic effects which may impact the perioperative course. As such, data are needed to clearly delineate the benefits of transfusion during the perioperative period.

DETAILED DESCRIPTION:
This prospective study will include patients presenting for spinal surgery. There will be no change in the anesthetic or perioperative care of these patients. Per our usual clinical routine, cell saver will be used intraoperatively to limit the need for allogeneic blood. Tissue and cerebral oxygenation will be monitored using near infrared spectroscopy (NIRS). The device is applied non-invasively like pulse oximetry to a muscle bed (usually the deltoid) and the forehead to measure tissue oxygenation. These devices are used routinely in the operating room and the cardiothoracic intensive care unit. Although not used on every major orthopedic procedure, these devices are routinely used in various high risk clinical scenarios. As clinically indicated, cell saver blood (autologous) or allogeneic blood will be administered. During this time, tissue and cerebral oxygenation will be recorded every 5 minutes starting 10 minutes before the transfusion and continued for 30 minutes following the transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing spinal surgery

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Spinal surgery patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-12; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Cerebral Oxygenation Changes | Intraoperative measure
  To evaluate changes in tissue and cerebral oxygenation during the administration of autologous or allogeneic blood during spinal surgery.

SECONDARY OUTCOMES:
Oxygenation Changes in Autologous versus Allogeneic Blood Transfusions | Intraoperative measure
  To determine if there are differences in the changes in tissue and cerebral oxygenation with autologous compared to allogeneic blood.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D. Tobias, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No